CLINICAL TRIAL: NCT03936426
Title: Peptide Receptor Radionuclide Therapy Administered to Participants With Meningioma With 67Cu-SARTATE™: A Single-centre, Open-label, Non- Randomised, Phase I-IIa Theranostic Clinical Trial
Brief Title: Peptide Receptor Radionuclide Therapy Administered to Participants With Meningioma With 67Cu-SARTATE™
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL02
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — 64Cu-SARTATE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARTATE (Experimental): All participants will receive 200 MBq of Cu-64 SARTATE given as a single bolus intravenous injection at Day 0. Participants will receive up to four administrations of Cu-67 SARTATE via a slow intravenous infusion over 30 minutes, 6 to 12 weeks apart. Individual activity administered per cycle will not exceed 5.1 GBq.
  Interventions: Drug: Cu-64 SARTATE and Cu-67 SARTATE

INTERVENTIONS:
Drug: Cu-64 SARTATE and Cu-67 SARTATE — Cu-64 SARTATE diagnostic drug Cu-67 SARTATE therapy drug
  Other Names: SARTATE; copper SARTATE; Cu-SARTATE; 64Cu-SARTATE; 67Cu-SARTATE; Cu-64 SARTATE; Cu-67 SARTATE; 64/67Cu-SARTATE; Cu-64/67 SARTATE

SUMMARY:
The primary purpose of this study is to investigate the safety and tolerability of a single dose of Cu-64 SARTATE and multiple doses of Cu-67 SARTATE administered to participants with meningioma. All participants in this study will be injected with a single dose of Cu-64 SARTATE to demonstrate how it is absorbed in the body. Then participants will receive individualised doses of Cu-67 SARTATE for up to 4 cycles.

DETAILED DESCRIPTION:
This is a single centre, open label, non-randomised, single cohort, multiple dose study of Cu-67 SARTATE administered to male and female participants diagnosed with grade I, II, or III meningioma. The maximum allowable dose will be calculated using dosimetry data acquired from PET/CT scans completed during a pre-treatment diagnostic & dosimetry phase using Cu-64 SARTATE, a structurally identical molecule radiolabelled with copper-64 (Cu-64), instead of copper-67 (Cu-67). Approximately 6 participants will be enrolled in the study. Participants will have up to 4 therapy cycles (6-12 weeks apart). Safety visits will occur between each cycle at bi-weekly intervals to ensure the participant meets the safety criteria prior to their next therapy. An efficacy assessment will be conducted following cycle 2 to determine if a subsequent 2 cycles of therapy will be administered. Participants who complete all four cycles of Cu-67 SARTATE therapy, will complete their final study visit at 12 weeks post administration of cycle 4.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age greater than or equal to 50 years.
3. Life expectancy greater than or equal to 3 months.
4. Has adequate organ function as defined by the following laboratory values obtained within 28 days prior to administration of Cu-64 SARTATE:

   1. Estimated glomerular filtration rate (eGFR) greater than 40ml/min as measured using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 3.0 x upper limit of normal (ULN).
   3. QT interval less than /=450msec as measured by 12 lead ECG.
5. Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2.
6. Diagnosis of recurrent or progressive histologically confirmed WHO grade I-III meningioma which has failed standard of care therapies. Patients will be considered to have failed standard care when they have disease that is progressing despite standard treatment (primarily radiotherapy) or where, in the opinion of their treating physician, further standard therapy is considered to be of sufficiently high risk of complication as to warrant consideration of alternate therapies.
7. Male participants must agree to use contraception methods from Day 0 through to 4 weeks after the last dose of Cu-67 SARTATE.
8. A female participant is eligible to participate if she is of:

   1. Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and oestradiol less than 40 pg/ml (less than 140 pmol/l) is confirmatory].
   2. Child-bearing potential and agrees to use contraception methods for an appropriate period of time (as determined by the Investigator) prior to Day 0 to sufficiently minimize the risk of pregnant females being enrolled. These measures are the combination of a barrier method AND established (greater than 2 cycles) hormonal methods (e.g. the oral contraceptive pill). Absolute sexual abstinence may be considered acceptable at the discretion of the investigator. Abstinence for the 12 days prior to therapy to allow for serum B-hCG assessment which should then ensure the patient is not pregnant prior to therapy administration.
   3. Female participants must agree to use contraception until four weeks after the last dose of Cu-67 SARTATE.

Exclusion Criteria:

1. Known sensitivity or allergy to somatostatin analogues.
2. Participants who have received interventional treatment for their meningioma within the four weeks prior to Day 0.
3. Any major surgery within the four weeks prior to Day 0.
4. Any additional planned interventions, including surgery or radiation therapy that would interfere with safety or efficacy assessments.
5. Treatment with long acting somatostatin analogues within 28 days prior to Day 0. Treatment with short acting somatostatin analogues within 24 hours prior to Day 0.
6. Any other malignancy in the past 5 years except for cervical intraepithelial neoplasia (CIN) of the cervix, squamous cell carcinoma (SCC) of the skin, basal cell carcinoma (BCC) of the skin or clinical insignificant prostate cancer not requiring prior therapy.
7. Breastfeeding females and pregnant females.
8. Treatment with any investigational agent received within four weeks prior to Day 0.
9. Participants unwilling or unable to comply with protocol requirements.
10. Urinary or faecal incontinence of sufficient degree to be of concern for contamination risk in the opinion of the Investigator.
11. Peptide receptor radionuclide therapy (PRRT) at any time prior to enrolment in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple doses of Cu-67 SARTATE using CTCAE version 4.03 | 55 weeks
  Safety will be assessed via vital signs, laboratory tests, physical examinations, ECGs and spontaneous adverse event reporting.
Safety and tolerability of a single dose of Cu-64 SARTATE using CTCAE version 4.03 | 56 weeks
  Safety will be assessed via vital signs, laboratory tests, physical examinations, ECGs and spontaneous adverse event reporting.

SECONDARY OUTCOMES:
Absorbed dose of Cu-64 SARTATE in target, non-target organs and whole body. | 1, 4 and 24 hours post administration of Cu-64 SARTATE.
  Absorbed doses (mSv/MBq) will be calculated using PET/CT scans acquired at 1, 4 and 24 hours post administration of Cu-64 SARTATE.
Absorbed dose of Cu-67 SARTATE in target, non-target organs and whole body. | 1, 4, 24 and 96 hours post administration of Cu-67 SARTATE.
  Absorbed doses (mSv/MBq) will be calculated using SPECT/CT scans acquired at 1, 4, 24 and 96 hours post administration of Cu-67 SARTATE.
Maximum and mean SUV of Cu-64 SARTATE in target organs and SSTR binding lesions. | 1, 4 and 24 hours post administration of Cu-64 SARTATE.
  Maximum and mean SUV will be calculated using PET/CT scans acquired at 1, 4 and 24 hours post administration of Cu-64 SARTATE.
Maximum and mean SUV of Cu-67 SARTATE in target organs and SSTR binding lesions. | 1, 4, 24 and 96 hours post administration of Cu-67 SARTATE.
  Maximum and mean SUV will be calculated using SPECT/CT scans acquired at 1, 4, 24 and 96 hours post administration of Cu-67 SARTATE.
Activity of Cu-64 SARTATE in target and non-target organs and SSTR binding lesions as a percentage of the administered dose. | 1, 4 and 24 hours post administration of Cu-64 SARTATE.
  The percentage of the administered dose will be calculated using PET/CT scans acquired at 1, 4 and 24 hours post administration of Cu-64 SARTATE.
Activity of Cu-67 SARTATE in target and non-target organs and SSTR binding lesions as a percentage of the administered dose. | 1, 4, 24 and 96 hours post administration of Cu-67 SARTATE.
  The percentage of the administered dose will be calculated using SPECT/CT scans acquired at 1, 4, 24 and 96 hours post administration of Cu-67 SARTATE.
Objective Response | At 6 weeks post second administration of Cu-67 SARTATE, as well as at 6 and 12 weeks following the fourth administration.
  Objective response to therapy will be assessed according to the RANO Response Criteria for Meningioma, as measured by MRI and clinical status.
Qualitative analysis of PET/CT scans post administration of Cu-64 SARTATE. | 1, 4 and 24 hours post administration of Cu-64 SARTATE.
  Qualitative analysis of PET/CT scans to identify uptake patterns.
Qualitative analysis of SPECT/CT scans post administration of Cu-67 SARTATE. | 1, 4, 24 and 96 hours post administration of Cu-67 SARTATE.
  Qualitative analysis of SPECT/CT scans to identify uptake patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Schembri, MD, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Royal North Shore Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bailey DL, Willowson KP, Harris M, Biggin C, Aslani A, Lengkeek NA, Stoner J, Eslick ME, Marquis H, Parker M, Roach PJ, Schembri GP. 64Cu Treatment Planning and 67Cu Therapy with Radiolabeled [64Cu/67Cu]MeCOSar-Octreotate in Subjects with Unresectable Multifocal Meningioma: Initial Results for Human Imaging, Safety, Biodistribution, and Radiation Dosimetry. J Nucl Med. 2023 May;64(5):704-710. doi: 10.2967/jnumed.122.264586. Epub 2022 Dec 2. PMID 36460344